CLINICAL TRIAL: NCT05340478
Title: Increasing the Effectiveness of CBT for Anxiety in Veterans by Involving Family Members.
Brief Title: Adjunctive Family CBT for Veterans With Anxiety
Acronym: AF-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3863-P
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorder
Keywords: panic; generalized anxiety; social anxiety; CBT
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Pilot feasibility trial with 2 phases. Phase 1 involved adapting and refining the AF-CBT intervention. Phase 2 involved a small pilot to assess feasibility of delivering the AF-CBT intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Initial) - Adapt/Refine AF-CBT (Other): Adjunctive Family - Cognitive Behavioral Therapy (AF-CBT) was adapted and refined for family members of Veterans with anxiety using an iterative process during Phase 1.
  Interventions: Behavioral: Adjunctive Family - Cognitive Behavioral Therapy
- Phase 2 (Final) - Pilot AF-CBT (Other): The final version of Adjunctive Family - Cognitive Behavioral Therapy (AF-CBT) was delivered to family members of Veterans with anxiety during Phase 2.
  Interventions: Behavioral: Adjunctive Family - Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Adjunctive Family - Cognitive Behavioral Therapy — AF-CBT provides family members psychoeducation on anxiety and teaches skills to facilitate the recovery of Veterans in the process of completing anxiety treatment.
  Other Names: AF-CBT

SUMMARY:
Despite the prevalence of posttraumatic stress disorder and anxiety disorders among Veterans, there has been limited focus on the development of interventions that include family members in treatments provided to Veterans. This is a feasibility study that examines a novel adjunct intervention (Adjunctive Family-Cognitive Behavioral Therapy; AF-CBT) developed for family members of Veterans undergoing behavioral treatment for anxiety-based disorders. Phase one involves piloting AF-CBT with family members and conducting qualitative interviews to obtain feedback about the utility and acceptability of the intervention. The refined protocol will be used in phase two, which involves an open trial where Veterans and family members will complete the intervention and attend a 1-month follow up assessment, including a qualitative interview.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) and anxiety disorders such as panic, generalized and social anxiety are highly prevalent among Veterans of all eras and negatively impact functioning and quality of life. Avoidance is a hallmark feature of anxiety and functions to maintain the disorder. Although cognitive behavior therapy (CBT) is effective, a significant proportion of Veterans show minimal improvement following treatment. This is often due to poor treatment adherence such as avoidance of using skills taught in CBT that require confronting distressing memories and feared situations. Avoidance behavior also can extend to caregivers and family members of Veterans, who may engage in accommodation behaviors (i.e., changing their own behaviors) to help alleviate distress experienced by their loved ones. As such, accommodation by family members undermines the effectiveness of CBT and is associated with greater symptom severity and functional impairment in persons with anxiety.

This study will examine the feasibility, acceptability, and satisfaction associated with a new intervention for family members of Veterans undergoing CBT for anxiety-based disorders. Adjunctive Family-CBT (AF-CBT) provides family members psychoeducation on anxiety and teaches skills that can be used to facilitate the recovery of Veterans who are in the process of completing treatment for anxiety. Aims of the study are to: (1) adapt and refine AF-CBT through an iterative process that will be informed by feedback from Veterans and family members; (2) examine the feasibility and acceptability/satisfaction of AF-CBT; (3) assess the validity and reliability of the Family Accommodation Scale-Anxiety adapted for Veterans and family members; and (4) examine the associations between family accommodation behavior and readjustment and anxiety in Veterans.

The proposed study involves a total of 47 Veterans and family member dyads (V/F dyad) and will be conducted in two phases. In phase 1, 12 V/F dyads will be recruited, and family members will receive AF-CBT while the Veteran undergoes iCBT for anxiety. The intervention will be delivered in three separate cohorts (approximately 4 V/F dyad in each cohort). During the 1-month assessment, information obtained from qualitative interviews will be used to refine the intervention in an iterative process with each cohort. In phase 2, 35 V/F dyads will be recruited and administered the finalized version of AF-CBT following the same treatment and assessment format. Qualitative interviews will focus on each V/F dyad's experience with the AF-CBT intervention and whether specific components of the intervention facilitated the Veteran's recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Veteran at least 18 years old;
* current diagnosis of at least one anxiety-based disorder: PTSD, PD, SAD, or GAD (based on ADIS-5);
* moderate-to-poor life enjoyment and satisfaction as indicated by a score of 47 or lower on the Q-LES-Q-SF
* BAI score of 16 (moderate anxiety) or higher;
* stable on psychotropic medication for 4 weeks before study participation; and
* has a family member willing to participate in the study

Exclusion Criteria:

* Active symptoms of mania or psychosis at baseline (based on ADIS-5);
* depression with active suicidal ideation/intent that would preclude treatment (based on ADIS-5 & BAI);
* moderate-to-severe cognitive impairment as indicated by a score below 20 on the SLUMS;
* active drug/alcohol abuse during the initial 3-months of study enrollment (otherwise Veterans with comorbid substance/alcohol dependence are study eligible); and
* undergoing concurrent transdiagnostic CBT for anxiety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred from Sept 2022 - Mar 2024 at the Michael E. DeBakey VA Medical Center.
Pre-assignment Details: There were a total of 7 dyads (14 participants comprised of 7 Veterans & 7 Family members) who were excluded after consenting (6 dyads did not meet inclusion criteria; 1 dyad was not clinically appropriate for the study).
Period: Overall Study
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
Started | 30 (Participants* eligible and enrolled in the study *15 Family Members; 15 Veterans) | 52 (Participant* eligible and enrolled in the study *26 Family Members; 26 Veterans)
Treatment Initiation | 21 (Participants* who initiated treatment (FM =AF-CBT; Veterans = iTCBT). *9 Family Members; 12 Veterans) | 48 (Participants* who initiated treatment (FM =AF-CBT; Veterans = iTCBT) *23 Family Members; 25 Veterans)
Treatment Completion | 15 (Participants* who completed treatment (FM =AF-CBT; Veterans = iTCBT). *7 Family Members; 8 Veterans) | 42 (Participants* who completed treatment (FM =AF-CBT; Veterans = iTCBT) *21 Family Members; 21 Veterans)
Completed Follow Up | 15 (Participants* who completed 1-month follow-up *7 Family Members; 8 Veterans) | 40 (Participants* who completed 1-month follow-up (FM=AF-CBT; Veterans = iTCBT). 20 Family Members; 20 Veterans)
Completed | 15 (Participants* who completed 1-month follow-up (FM =AF-CBT; Veterans = iTCBT). *7 Family Members; 8 Veterans) | 40 (Participants who completed 1-month follow-up. Note: Follow-up data were collected from 20 Veterans and 20 Family Members.)
Not Completed | 15 | 12
Not completed — Scheduling Issues | 10 | 4
Not completed — Neither member of dyad started treatment | 2 | 2
Not completed — Withdrawn from study | 2 | 2
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Population: Phase 1 included 8 dyads (8 Family Members; 8 Veterans). Phase 2 included 21 dyads (21 Family Members; 21 Veterans). This only includes dyads who initiated treatment and have follow-up data.
  Note: The following data were not collected from family members: Age & BAI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT | Total
Number analyzed (Participants) | 16 | 42 | 58
Age, Categorical [Count of Participants; unit: Participants] — These data are only available for Veteran participants. Population: These data were only collected from Veterans. This information was not collected from Family Members.
  Participants
    number analyzed (Participants) | 8 | 21 | 29
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 7 | 21 | 28
    >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: These numbers represent data collected from Veterans only. This data was not collected from Family Members.
  years
    number analyzed (Participants) | 8 | 21 | 29
    (all) | 48.13 (13.35) | 45.62 (11.47) | 46.31 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed includes individual participants (Veterans & Family Members)
  Participants
    Veterans: number analyzed (Participants) | 8 | 21 | 29
    Veterans: Female | 1 | 4 | 5
    Veterans: Male | 7 | 17 | 24
    Family Members: number analyzed (Participants) | 8 | 21 | 29
    Family Members: Female | 7 | 16 | 23
    Family Members: Male | 1 | 5 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall count of 16 in Phase 1 includes data from 8 Veterans and 8 Family Members. The overall count of 42 in Phase 2 includes data from 21 Veterans and 21 Family Members.
  Participants
    Veterans: number analyzed (Participants) | 8 | 21 | 29
    Veterans: Hispanic or Latino | 1 | 6 | 7
    Veterans: Not Hispanic or Latino | 7 | 15 | 22
    Veterans: Unknown or Not Reported | 0 | 0 | 0
    Family Members: number analyzed (Participants) | 8 | 21 | 29
    Family Members: Hispanic or Latino | 3 | 8 | 11
    Family Members: Not Hispanic or Latino | 5 | 12 | 17
    Family Members: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: For Phase 1 the total count of 16 participants includes 8 Veterans and 8 Family Members. For Phase 2 the total count of 42 participants includes 21 Veterans and 21 Family Members.
  Participants
    Veteran: number analyzed (Participants) | 8 | 21 | 29
    Veteran: American Indian or Alaska Native | 0 | 0 | 0
    Veteran: Asian | 1 | 0 | 1
    Veteran: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Veteran: Black or African American | 0 | 3 | 3
    Veteran: White | 4 | 15 | 19
    Veteran: More than one race | 3 | 1 | 4
    Veteran: Unknown or Not Reported | 0 | 2 | 2
    Family Member: number analyzed (Participants) | 8 | 21 | 29
    Family Member: American Indian or Alaska Native | 0 | 0 | 0
    Family Member: Asian | 1 | 0 | 1
    Family Member: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Family Member: Black or African American | 1 | 3 | 4
    Family Member: White | 5 | 10 | 15
    Family Member: More than one race | 0 | 5 | 5
    Family Member: Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 42 | 58

OUTCOME MEASURES:

1. Primary Outcome: Modified Treatment Evaluation Inventory
Description: Degree to which treatment components were found to be acceptable. Scores range from 9-45, with higher scores reflecting greater acceptance of treatment.
Time Frame: 1-month follow-up
Population: In Phase 1, 1 family member did not complete this measure. In Phase 2, 1 Veteran and 2 Family Members did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
Number analyzed (Participants) | 15 | 39
score on a scale
  Veteran: number analyzed (Participants) | 8 | 20
  Veteran | 32.13 (3.31) | 35.40 (5.11)
  Family Member: number analyzed (Participants) | 7 | 19
  Family Member | 34.29 (4.07) | 35.32 (4.73)

2. Primary Outcome: Client Satisfaction Questionnaire
Description: Degree to which participant was satisfied with treatment. Scores range from 8-32, with higher scores reflecting greater satisfaction.
Time Frame: 1-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
Number analyzed (Participants) | 15 | 39
score on a scale
  Veteran: number analyzed (Participants) | 8 | 20
  Veteran | 26.63 (3.16) | 28.60 (3.62)
  Family Member: number analyzed (Participants) | 7 | 19
  Family Member | 27.00 (3.16) | 28.42 (3.66)

3. Primary Outcome: Feasibility of Recruitment for AF-CBT
Description: This outcome pertains to the feasibility of recruiting participant dyads for the AF-CBT intervention across Phases 1 and 2 of the study. The rate of recruitment is based on the number of dyads who agreed to participate out of those invited during the active recruitment period for this study.
Time Frame: Recruitment Initiation to Recruitment Completion (up to 18 Months)
Population: A total of 64 dyads (Veterans & Family Members) were invited to participate in the study.
Measure: Number; unit: dyads
Groups:
- AF-CBT: Adjunctive Family -CBT for family members of Veterans with anxiety
  Intensive Transdiagnostic Cognitive Behavioral Therapy: cognitive behavioral treatment that addresses multiple anxiety problems simultaneously and delivered in a massed format over one weekend
Arm/Group | AF-CBT
Number analyzed (Participants) | 64
dyads | 48

4. Secondary Outcome: Beck Anxiety Inventory
Description: Measure of anxiety including cognitive and somatic components of anxiety. Scores range from 0-63, with higher scores reflecting higher levels of anxiety.
  Note: The BAI was not collected from family members.
Time Frame: Baseline; 1-Month Follow-Up
Population: One Veteran in Phase 2 did not complete the BAI at the 1-Month Follow-Up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
Number analyzed (Participants) | 8 | 21
score on a scale
  Baseline Veteran | 35.00 (11.20) | 32.62 (11.74)
  1 Month Veteran: number analyzed (Participants) | 8 | 20
  1 Month Veteran | 31.25 (17.25) | 19.20 (12.63)
Statistical Analysis 1: Comparison: Phase 1 (Initial) - Adapt/Refine AF-CBT vs Phase 2 (Final) - Pilot AF-CBT; Test type: Superiority; p < .001, t-test, 2 sided

5. Secondary Outcome: Family Accommodation Scale
Description: Degree to which family member engages in accommodation behaviors. Scores range from 0-36, with higher scores reflecting greater levels of accommodation.
Time Frame: Baseline; 1-Month Follow-Up
Population: In Phase 1, 1 family member did not complete this measure at the 1-month follow-up. In Phase 2, 1 Veteran and 2 Family Members did not complete this measure at the 1-month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
Number analyzed (Participants) | 16 | 42
units on a scale
  Baseline Family Member: number analyzed (Participants) | 8 | 21
  Baseline Family Member | 21.75 (8.45) | 19.86 (8.51)
  1 Month Family Member: number analyzed (Participants) | 7 | 19
  1 Month Family Member | 25.00 (7.83) | 15.05 (7.60)
  Baseline Veteran: number analyzed (Participants) | 8 | 21
  Baseline Veteran | 20.50 (9.07) | 19.62 (9.21)
  1 Month Veteran: number analyzed (Participants) | 8 | 20
  1 Month Veteran | 19.75 (8.14) | 18.00 (9.41)

6. Primary Outcome: Feasibility of Retention for AF-CBT
Description: This outcome pertains to the feasibility of retaining participant dyads for the AF-CBT intervention across Phases 1 and 2 of the study. The rate of retention is the percentage of dyads who complete AF-CBT by attending all sessions.
Time Frame: Baseline to Treatment Completion (average 4 months)
Population: In Phase 1, of the 30 participants (Veterans & Family Members) enrolled, 15 completed treatment. In Phase 2, of the 52 participants (Veterans & Family Members) enrolled, 39 completed treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
Number analyzed (Participants) | 30 | 52
Participants | 15 | 39

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 5 months.
Description: Note: Adverse events were not collected from family members.
Arm/Group | Phase 1 (Initial) - Adapt/Refine AF-CBT | Phase 2 (Final) - Pilot AF-CBT
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/21
Other Adverse Events (participants affected / at risk) | 0/8 | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Initial) - Adapt/Refine AF-CBT (N=8) | Phase 2 (Final) - Pilot AF-CBT (N=21)
Visit to ER (General disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT05340478/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT05340478/ICF_000.pdf